CLINICAL TRIAL: NCT06409936
Title: Asciminib as Single Agent or in Combination With Nilotinib in the 1st-line Treatment of BCR-ABL1+ Chronic Myeloid Leukemia: a Randomized GIMEMA-GELMC Phase II Study PEARL Study: PotEntial of Asciminib in the eaRly Treatment of CML
Brief Title: PEARL Study: PotEntial of Asciminib in the eaRly Treatment of CML
Acronym: PEARL
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Gruppo Italiano Malattie EMatologiche dell'Adulto (Other)
Collaborators: Grupo Español de Leucemia Mieloide Crónica (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CML1624
Record Dates: First submitted 2024-05-07; First posted 2024-05-10 (Actual); Last update posted 2025-07-08 (Actual); Status verified 2025-07

CONDITIONS: CML, Chronic Phase; Chronic Myeloid Leukemia, Chronic Phase; Chronic Myeloid Leukemia, BCR/ABL-Positive; Chronic Myeloid Leukemia
Keywords: asciminib; nilotinib
MeSH Terms: conditions — Leukemia, Myeloid, Chronic-Phase; Leukemia, Myelogenous, Chronic, BCR-ABL Positive | interventions — asciminib; nilotinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Asciminib single agent (Experimental): Core phase (2 years): asciminib 80 mg QD will be given as single-agent.
  Consolidation phase (2 years): If patients will have achieved a DMR (MR4), or if it will be in their interest, the treatment will be continued with asciminib 80 mg QD.
  Treatment free remission phase (1 year): patients maintaining a stable MR4 up to the end of the fourth year will discontinue the treatment
  Interventions: Drug: Asciminib
- Asciminib plus nilotinib (Experimental): Core phase (2 years): asciminib 80 mg QD will be started, then after 90 days asciminib will be given 40 mg BID and nilotinib 300 mg BID, or 300 mg OAD according to the presence/absence of asciminib adverse events, will be added-on.
  Consolidation phase (2 years): If patients will have achieved a DMR (MR4), or if it will be in their interest, the treatment will be continued with asciminib 40 mg BID and nilotinib reduced to 300 mg daily.
  Treatment free remission phase (1 year): patients maintaining a stable MR4 up to the end of the fourth year will discontinue the treatment
  Interventions: Drug: Asciminib; Drug: Nilotinib

INTERVENTIONS:
Drug: Asciminib — both arms will include asciminib treatment
Drug: Nilotinib — in the arm B the nilotinib will be added on in all patients
  Arms: Asciminib plus nilotinib

SUMMARY:
A phase 2, interventional, randomized unblinded study will be conducted in newly diagnosed CP CML patients, to investigate the efficacy and the safety of asciminib at a dose of 80 mg QD as single agent (arm A) or 40 mg BID in combination with nilotinib 300 mg BID (arm B).

All patients in both arm A and arm B will be treated for a minimum of 2 years (core phase). If they will have achieved a DMR (MR4), or if it will be in the interest of the patient, the treatment will be continued.

During the consolidation phase (2 years) asciminib will be continued at the same dose in both arms; in the combination arm the nilotinib dose will be reduced to 300 mg daily.

The patients maintaining a stable MR4 up to the end of the fourth year will discontinue the treatment (TFR phase). The rate of TFR at 5 year (1 year after discontinuation) will be evaluated.

DETAILED DESCRIPTION:
A phase 2, prospective, interventional, randomized (two arms, randomization 1:1), unblinded study will be conducted in newly diagnosed CP CML patients, to investigate the efficacy and the safety of asciminib at a dose of 80 mg QD as single agent (arm A) or 40 mg BID in combination with nilotinib 300 mg BID (arm B).

* In the arm A, asciminib 80 mg QD will be given as single-agent. In the arm B, asciminib 80 mg QD will be started, then after 90 days asciminib will be given 40 mg BID and nilotinib 300 mg BID, or 300 mg OAD according to the presence/absence of asciminib adverse events, will be added-on in all patients. All patients in both arm A and arm B will be treated for a minimum of 2 years (core phase). If they will have achieved a DMR (MR4), or if it will be in the interest of the patient, the treatment will be continued. In both arms the study drugs may be discontinued at any time for inefficacy (failure) or safety reasons(grade 3-4 toxicity or persistent grade 2 non hematologic toxicity). However, all the patient will remain "in study" (regular follow-up information will be required). The dose adjustments for toxicity and detailed criteria for treatment discontinuation (asciminib in arm A; asciminib or nilotinib in arm B) are specified within the protocol.
* After the induction of a DMR, the residual disease will be closely monitored by Q-PCR until the fourth year (consolidation phase). During the consolidation phase (2 years) asciminib will be continued at the same dose in both arms; in the combination arm the nilotinib dose will be reduced to 300 mg daily.
* The patients maintaining a stable MR4 up to the end of the fourth year, that must include in the last year at least 3 evaluable QPCR analyses, will enter the treatment free remission (TFR) phase of the study and will discontinue the treatment (TFR phase). A single unconfirmed loss of MR4 will not preclude the possibility of treatment discontinuation. In case of confirmed loss of MR3 after discontinuation, the choice of subsequent treatment will be up to Local Investigators. The rate of TFR at 5 year (1 year after discontinuation) will be evaluated.

ELIGIBILITY:
Inclusion Criteria:

* Cytogenetic and molecular confirmed diagnosis of Ph+ and BCR::ABL1+ CML
* Age ≥ 18 years
* Early chronic phase, less than 3 months from diagnosis
* Evidence at the time of study entry of typical BCR::ABL1 RNA transcripts e13a2 or e14a2 (b2a2 or b3a2), which are required for BCR::ABL1 international scale reporting
* Prior treatment with any TKI for 30 days or less; prior treatment with hydroxyurea or anagrelide is allowed
* ECOG performance status of 0, 1 or 2
* Adequate end organ function as defined by Total bilirubin ≤ 1.5 x ULN except for patients with Gilbert's syndrome who may only be included if total bilirubin ≤ 3.0 x ULN or direct bilirubin ≤ 1.5 x ULN Aspartate transaminase (AST) ≤ 3.0 x ULN Alanine transaminase (ALT) ≤ 3.0 x ULN Serum amylase ≤ ULN Serum lipase ≤ ULN Alkaline phosphatase ≤ 2.5 x ULN, unless considered tumor related Creatinine clearance > 50 ml/min using Cockcroft-Gault formula
* Signed written informed consent according to ICH/EU/GCP and national local laws prior to any study procedure
* An effective form of contraception with their sexual partners from enrolment through 30 days after the end of treatment

Exclusion Criteria:

* CML in blast phase (BP) or in second chronic phase after previous BP, according to WHO criteria
* Previous treatment with TKIs for more than 30 days
* Refusal or impossibility to give an informed consent
* History or current diagnosis of cardiac disease indicating significant risk of safety for patients participating in the study such as uncontrolled or significant cardiac disease, including any of the following: recent myocardial infarction (within last 6 months), uncontrolled congestive heart failure, unstable angina (within last 6 months), clinically significant (symptomatic) cardiac arrhythmias (e.g., sustained ventricular tachycardia, and clinically significant second or third degree AV block without a pacemaker).
* Severe and/or uncontrolled concurrent medical disease that in the opinion of the investigator could cause unacceptable safety risks or compromise compliance with the protocol (e.g. uncontrolled diabetes, active or uncontrolled infection)
* History of acute pancreatitis within 1 year of study entry or past medical history of chronic pancreatitis
* History of acute or chronic liver disease
* History of other active malignancy within 2 years prior to study entry with the exception of previous or concomitant basal cell skin cancer and previous carcinoma in situ treated curatively
* Known history of Human Immunodeficiency Virus (HIV), Hepatitis B (HBV), or Hepatitis C (HCV) infection. Testing for Hepatitis B surface antigen (HBs Ag) and Hepatitis B core antibody (HBc Ab / anti HBc) will be performed at study entry
* Impairment of gastrointestinal (GI) function or GI disease that may significantly alter the absorption of study drug (e.g. ulcerative disease, uncontrolled nausea, vomiting, diarrhea, malabsorption syndrome, small bowel resection, or gastric bypass surgery)
* Pregnant or lactating women, where pregnancy is defined as the state of a female after conception and until the termination of gestation, confirmed by a positive hCG laboratory test.
* Women of child-bearing potential, unless they are using highly effective methods of contraception during dosing and for 30 days after the end of treatment

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 160 (Estimated)
Dates: Start 2025-06-26 (Actual); Primary Completion 2029-06 (Estimated); Study Completion 2032-06 (Estimated)

PRIMARY OUTCOMES:
evaluation of response of asciminib single-agent or in combination with nilotinib | at 2 years
  Rate of deep molecular response (MR4) achievement

CONTACTS AND LOCATIONS:
Overall Officials: Fausto Castagnetti, Principal Investigator — "Seragnoli" Institute of Hematology Bologna (Italy); Valentin Garcia Gutierrez, Principal Investigator — Hematology Unit, Hospital Universitario Ramón y Cajal, Madrid (Spain)
Locations (11):
- Spain (11):
  - Hospital del Mar (Barcelona), Barcelona
  - Hospital Universitario Basurto, Bilbao
  - Institut Català d'Oncologia Girona, Girona
  - Hospital Virgen de las Nieves, Granada
  - Hospital Universitario de Gran Canaria Dr. Negrín, Las Palmas de Gran Canaria
  - Hospital Gral U. Gregorio Marañón, Madrid
  - Hospital Universitario 12 de Octubre, Madrid
  - Hospital Universitario La Paz, Madrid
  - Hospital Clínico Universitario Virgen de la Arrixaca, Murcia
  - Complejo Asistencial Universitario de Salamanca, Salamanca
  - Hospital Universitario La Fe Valencia, Valencia